CLINICAL TRIAL: NCT00773227
Title: Treatment of Dysphagia in Oculopharyngeal Muscular Dystrophy by Autologous Transplantation of Myoblasts
Acronym: OPMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P020908; AOM02100
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Muscular Dystrophy, Oculopharyngeal
Keywords: Oculopharyngeal muscular dystrophy; Swallowing disorders, dysphagia; Pharyngeal propulsion; Upper oesophageal sphincter; Cricopharyngeal muscle; Autologous myoblasts; Autograft; Myotomy of the upper oesophageal sphincter; Fibroscopy of swallowing; Videofluoroscopy of swallowing
MeSH Terms: conditions — Muscular Dystrophy, Oculopharyngeal; Deglutition Disorders | interventions — Myotomy; Transplantation, Autologous; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All patients included
  Interventions: Procedure: Autologous myoblasts transplantation and myotomy

INTERVENTIONS:
Procedure: Autologous myoblasts transplantation and myotomy — Graft of autologous cell muscles (myoblasts) isolated from unaffected limb muscles into the pharyngeal muscles of patients diagnosed as suffering from OPMD and surgical procedure (myotomy)
  Other Names: autograft and surgery

SUMMARY:
The OCULO-Pharyngeal Muscular Dystrophy (OPMD) is a late onset hereditary muscle disease which is characterised by the selective affection of the pharyngeal muscles resulting in swallowing disorders, and by a ptosis from the dysfunction of the levator palpebral superiors muscles. Swallowing disorders are determinant in the prognosis of the disease, and potentially life-threatening deglutition, due to aspiration and denutrition. Degenerative dystrophy of the pharyngeal muscles causes difficulties to prepulse the food bolus in the pharynx, and the decreased relaxation of the cricopharyngeal muscle induced by the disease leads to blockage of food in the upper esophageal sphincter. The most common treatment for the dysphagia in OPMD is a myotomy of the upper esophageal sphincter muscles. However, although this will relax the constriction of the upper esophageal sphincter muscles and improve transitory the swallowing, it will not prevent the progressive degradation of the pharyngeal muscles. This progressive loss of contractility will eventually result in aspiration and severe difficulty in swallowing, increasing risk of aspiration pneumonia and severe weight loss which are the most common causes of mortality in OPMD patients.

The protocol which we are proposing is a graft of autologous cell muscles (myoblasts) isolated from unaffected limb muscles into the pharyngeal muscles of patients diagnosed as suffering from OPMD. Our aim is to improve both swallowing and the contractile deficit generated by the dystrophic pharyngeal muscles. A myotomy of the upper esophageal sphincter will be carried out at the same time as the myoblast transplantation, since we have already validated the improvement resulting from this surgery. Advantages of this new therapy in OPMD is the autograft, without risks of rejection, and the graft of myoblasts into the dystrophic pharyngeal muscles, above the myotomy of the upper esophageal sphincter muscles.

This model of cellular therapy has been studied through a preclinical study performed in dogs, allowing to valid the procedure and its safety, as well as to study the survival myoblasts grafted in the pharyngeal muscles.

This protocol is proposed for OPMD patients; it is firstly a safety study of both autograft and surgical procedure. In addition, the autograft may improve the swallowing disorders and life-threatening complications induced by aspiration and weight loss, resulting in a potential individual benefit.

DETAILED DESCRIPTION:
OCULO-Pharyngeal Muscular Dystrophy (OPMD) is characterised by the selective affection of the superior sphincter muscles of the oesophagus (SSO) and the pharyngeal.muscles resulting in dysphagia. The most common treatment for the dysphagia induced by this disease is a myotomy. However, although this will relax the constriction and improve swallowing it will not prevent the progressive degradation of the pharyngeal muscles. This progressive loss of contractility will eventually result in false routes and severe difficulty in swallowing, increased risk of pulmonary infection and severe weight loss which are the most common causes of mortality in these patients.

Concept:

The protocol which we are proposing is a pilot study in which autologous myoblasts isolated from unaffected limb muscles will be grafted into the pharyngeal constrictor muscles of patients diagnosed as suffering from OPMD. Our aim is to improve both swallowing and the contractile deficit generated by the dystrophic pharyngeal constrictor muscles. A myotomy of the SSO will be carried out at the same time as the myoblast transplantation, since we have already validated the improvement resulting from this surgery even though we know that this will provide only a partial and transitory improvement.

Type of trial: This is a multicentric trial with a direct benefit for the patient in which 10 patients will receive an autologous transplantation of myoblasts. Due to the possibility that a certain number of patients may withdraw from the study we have decided to include initially a maximum of 15 patients. The PHRC for this clinical trial was accepted in 2002 and the official promotor is the AP-HP. The patients will be selected by the different promotors but will be followed in the 'Service d'ORL of TENON Hospital '. The proliferative capacity of the myoblasts isolated from the muscle biopsies will be carried out by Vincent MOULY and KAMEL MANCHAOUI in the UMR 7000 CNRS directed by Dr Butler-Browne and the cells will be amplified prior to grafting in the Cellular laboratory therapy of Dr MAROLLEAU; The clinical trial will be controlled by a specifically selected committee of five.

Description of the trial In the first step of this study patients will be selected for inclusion in the trial according to the following criteria : 1: men or women aged between 18 and 75 years ; 2: genetic confirmation and characterisation of OPMD 3: SSO dysfunction confirmed by the stasis of saliva or food above the sphincter visualised by fibroscopy and a defect in the opening of the SSO also confirmed by videofluoroscopy of swallowing; the SSO defect may be associated with a reduction in pharyngeal propulsion as revealed by fibroscopy and videofluoroscopy of swallowing 4: official signed consent of the patients to participate in this clinical trial.

The next step will be the selection of the unaffected muscle to be used for the production of the autologous myoblasts to be used for transplantation. Muscles will be selected for engraftment on the basis of the proliferative capacity of the cultures made from biopsies (0.5-1gm) obtained following local anesthesia of either the quadriceps or the STERNO-CLEIDO-MASTOIDIEN muscles. The muscle which is able to produce the largest number of myoblasts will be biopsied a second time using the same conditions. Two grams of muscle will be removed and the myoblasts will be isolated and cultured until there are about 100 million myoblasts at which point the cells can be injected into the pharyngeal muscles of the patient. If there is no difference between the two different muscle biopsies then we will biopsy preferentially the STERNO-CLEIDO-MASTOIDIEN muscle since it is situated directly in the trajectory that will be used when grafting the myoblasts. The operation by lateral cervicotomy will be carried out under general anesthesia, in order to expose the SSO and the pharyngeal muscles. The graft will be carried out by injecting the myoblasts into about 20 different sites in the pharyngeal constrictor muscles above the site of the associated myotomy of the SSO. The next step will involve a two year evaluation of the trial. For each patient a descriptive analysis will be carried out based on the comparison of the different results. The principal evaluation of the efficiency of the graft will be based on the functional quality of the pharyngeal propulsion as determined by fibroscopy and videofluoroscopy of swallowing. A secondary evaluation will be based on the global swallowing properties which will be evaluated by a quantitative test, by a questionnaire and by an evaluation of the tolerance. This evaluation will include a clinical examination at each visit consisting of the examination of the pharynx in order to confirm the absence of muscle tumors and a cervical palpation in order to determine the volume of the muscle and to survey the site of myoblasts implantation. A rigid tube pharyngeal endoscopy which will be carried out under general anesthesia 6 to 12 months after the graft in case of abnormal pharynx at fibroscopy. In addition, a global neuromuscular examination will be carried out on an annual basis to follow the general evolution of the myopathy. The fibroscopy to determine the swallowing function, the global quantitative tesy of swallowing and the questionnaire will be carried out at 2, 6 and 24 months after the graft. A videofluoroscopy of swallowing will be carried out at 2 months then at 1 and 2 years after the graft.

Risks and Benefits:

The principal benefits to the patients which could be envisioned by this procedure is a delay in the deterioration of the pharyngeal muscles associated with this disease and consequently an improvement in the difficulties in swallowing usually associated with this disease. The potential risk associated with this type of operation are an inflammatory reaction, the appearance of a tumor or the lack of improvement of the symptoms associated with the disease.

A parallel preclinical study has been carried out in the dog in order to evaluate the tolerance and feasibility of the procedure for autografting myoblasts in the pharyngeal muscles.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman <18-75> years old
* Oculopharyngeal muscular dystrophy confirmed by genetic diagnosis (mutation of the GCG) on the chromosome 14)
* Oculopharyngeal muscular dystrophy with UES dysfunction

  1. salivary or alimentary stasis at fibroscopy of swallowing above the UES,
  2. decreased opening of the UES at videofluoroscopy of swallowing A decreased of the pharyngeal propulsion may be associated Written consent of the patient

Exclusion Criteria:

* History of myotomy of the UES in the context of the Oculopharyngeal muscular
* Dystrophy;
* HIV, hepatitis B or C tuberculosis);
* Lupus, rheumatoid polyarthritis, sarcoïdosis, collagenosis) ;
* Other neuromuscular diseases ;
* History of malignant tumor ;
* History of neck radiotherapy ;
* Renal failure (creatinine clearance <60ml/min)
* Liver failure ;
* Pregnancy ;
* Follow up less than 24 months:
* Patients who refuse to sign the consent;
* No social security.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-04; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The principal evaluation of the efficiency of the graft will be based on the functional quality of the pharyngeal propulsion as determined by fibroscopy and videofluoroscopy of swallowing. | before the graft and at 2, 6, 12, 18 and 24 months after the graft

SECONDARY OUTCOMES:
on the global swallowing properties which will be evaluated by a quantitative test, by a questionnaire and by an evaluation of the tolerance. This evaluation will include a clinical examination at each visit consisting | before the graft and at 2, 6, 12, 18 and 24 months after the graft

CONTACTS AND LOCATIONS:
Overall Officials: Jean Lacau-Saint Guily, MD, PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hospital Tenon, Paris, France

REFERENCES:
- [Derived] Perie S, Trollet C, Mouly V, Vanneaux V, Mamchaoui K, Bouazza B, Marolleau JP, Laforet P, Chapon F, Eymard B, Butler-Browne G, Larghero J, St Guily JL. Autologous myoblast transplantation for oculopharyngeal muscular dystrophy: a phase I/IIa clinical study. Mol Ther. 2014 Jan;22(1):219-25. doi: 10.1038/mt.2013.155. Epub 2013 Jul 8. PMID 23831596